CLINICAL TRIAL: NCT04951414
Title: Study on the Rehabilitation Treatment of Knee Osteoarthritis Based on ICF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: D181100000318004
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICF
  Interventions: Diagnostic Test: ICF core set
- Control

INTERVENTIONS:
Diagnostic Test: ICF core set — KOA rehabilitation regimen based on the complete core combination of ICF was accepted
  Groups: ICF

SUMMARY:
To solve the existing Knee osteoarthritis;KOA) clinical norms and guidelines have low operability, Disconnection between treatment plan and specific evaluation results, difficulty in achieving individualized intervention and other problems, on the one hand, we need to develop Chinese expert consensus or clinical path based on evidence-based medicine to adapt to China's national conditions, on the other hand, is more important in The KOA clinical process introduces a set of tools to translate evidence-based medicine evidence into specific, actionable treatments, Thus, a more flexible, more comprehensive and three-dimensional, adaptable, targeted, more conducive to the promotion of the individual integration KOA rehabilitation intervention program.

ELIGIBILITY:
Inclusion Criteria:

* Neither knee had undergone knee replacement, and no knee replacement had been performed in recent half a year planning to have a knee replacement; Volunteered to participate in the study and signed the informed consent.

Exclusion Criteria:

* People with consciousness disorder, cognitive disorder, severe mental illness, unable to accurately express their own will, or unable to cooperate with the completion of various assessments and treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Six hundred patients with knee osteoarthritis were treated in each participating research unit
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
treatment compliance | 1month
  treatment compliance of rehabilitation treatment
treatment compliance | 3month
  treatment compliance of rehabilitation treatment
treatment compliance | 6month
  treatment compliance of rehabilitation treatment

CONTACTS AND LOCATIONS:
Overall Officials: YUANMINGFEI ZHANG, Study Director — Peking University Third Hospital
Locations (2):
- China (2):
  - Capital clinical characteristic applied research and achievement promotion, Beijing, Beijing Municipality
  - Huarunwugang general hospital, Wuhan, Hubei